CLINICAL TRIAL: NCT00997412
Title: Randomized, Double-blind, Double-dummy Trial of Mycophenolic Acid Versus Azathioprine in the Treatment of Corticosteroid-refractory Myasthenia Gravis
Brief Title: Trial of Mycophenolic Acid Versus Azathioprine in the Treatment of Corticosteroid-refractory Myasthenia Gravis
Acronym: Myfortic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qualitix Clinical Research Co., Ltd. (Industry)
Responsible Party: Jiann-Horng Yeh / M.D., Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CERL080ATW07T
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MA (Experimental): MA group: 1 tablet AZA placebo and 4 tablets MA (180mg/tab,720 mg/day) twice daily
  Interventions: Drug: Mycophenolic acid
- AZA (Active Comparator): AZA group: 1 tablet AZA (50mg/tab) and 4 tablets MA placebo twice daily
  Interventions: Drug: AZA

INTERVENTIONS:
Drug: Mycophenolic acid — 180 mg/tablet, 4 tablets twice daily
  Arms: MA
Drug: AZA — 1 tablet AZA (50 mg/tab) and 4 tablets MA placebo twice daily
  Arms: AZA

SUMMARY:
This is an randomized, double-blind, double-dummy trial, and the objective is to compare the efficacy and safety of Mycophenolic acid (MA) and Azathioprine (AZA), immunosuppressive drugs, in myasthenia gravis patients. This prospective study will enroll 40 myasthenia gravis (MG) patients who are poor controlled under prior steroid therapy. All subjects should be randomly assigned to MA group and AZA group that will receive routine pyridostigmine and prednisolone in combination with MA or AZA.

DETAILED DESCRIPTION:
This will be a double-dummy study to keep the blinded quality.

* MA group: 1 tablet AZA placebo and 4 tables MA (180 mg/tab,720 mg/day) twice daily.
* AZA group: 1 tablet AZA (50mg/tab) and 4 tables MA placebo twice daily.

  * When patients achieve minimal manifestation (MM, i.e. complete remission), which lead to normal daily routine, the dose of pyridostigmine should reduce to 240 mg/day (4 tablets) or less. The dose of steroid should be stepped down by 10 mg qod (every other day) for every 2 weeks until the dose achieves 40 mg qod. After that, the dose should be stepped down by 5 mg qod for every month.
  * When disease progresses and is no longer maintaining minimal manifestation, the dose of steroid will be stepped up by 10 mg qod for every 2 weeks until achieve clinical stable remission. The taper rule of steroid could start again 1 month after stabilization.
  * Every patient will be treated for 1 year. If the patient could not achieve MM within 1 year, the blind of individual patient will be opened and the patients will be crossed over to another medical treatment. The efficacy and safety of second medication will be observed openly until the end of study.
  * When the muscle weakness worsens under established study schedule, plasmapheresis could be conducted to improve the condition rapidly.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age between 20-70 (including 20 and 70 years old).
* Osserman II and III Myasthenia Gravis.
* Positive serum anti-acetylcholine receptor antibodies.
* Poor control of disease with daily dose of prednisone ≥ 30 mg or 0.5 mg/kg at 3 months before enrollment.
* Without immunosuppressive therapy other than steroid.

Exclusion Criteria:

* Ocular MG or minimal clinical syndrome that would not require the therapy of steroids.
* Negative serum anti-acetylcholine receptor antibodies.
* Use immunosuppressants other than steroids in the preceding year.
* Previous use other investigational medication within 3 months or current participate other clinical study.
* Poor renal function: serum creatinine > 3.0 mg/dl or estimated creatinine clearance < 30 ml/min
* Females who are pregnancy or breast-feeding.
* Recent history, within 5 years, of malignancy
* Unwilling or unable to participate the necessary continuous visits and examinations.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
The ratio of two arms patients achieve minimal manifestation (MM, i.e. complete remission) | One year after treatment

SECONDARY OUTCOMES:
Osserman clinical classification | One year after treatment
Myasthenia gravis (MG) score | One year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jiann-Horng Yeh, M.D., Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital